CLINICAL TRIAL: NCT06325904
Title: Uniportal Video Assisted Thoracoscopic Surgery (VATS) Debridement Versus Chest Tube Drainage in Early Stage Empyema
Brief Title: Uniportal VATS Versus Chest Tube for Early Empyema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Yasser Ali Kamal, Clinical professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9138930
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Empyema, Pleural
Keywords: Video-assisted thoracoscopic surgery; Pleura; Empyema
MeSH Terms: conditions — Empyema, Pleural; Empyema | interventions — Chest Tubes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): * This group included 30 adult patients with stage I/II pleural empyema who operated initially by VATS.
  * All patients were subjected to the following:
    1. Full history taking. 2.Full clinical examination. 3-Routine Laboratory investigations and Pleural fluid sample analysis. 4- Radiological investigations: Chest X-ray , CT chest.
  * All patients will be managed by general anesthesia using double lumen endoteracheal tube to achieve single lung ventilation.
  * All patients were positioned in lateral decubitus position.
  * Single port skin incisions was made to pass the port through which the camera head and instruments were introduced into the chest .
  * One chest tubes ws inserted as drains.
  Interventions: Procedure: Uniportal VATS
- 2 (Placebo Comparator): * This group included 30 adult patients with stage I/II pleural empyema who underwent conventional tube thoracotomy.
  * All patients were subjected to the following:
    1. Full history taking. 2.Full clinical examination. 3-Routine Laboratory investigations and Pleural fluid sample analysis. 4- Radiological investigations: Chest X-ray , CT chest.
  * The patient is placed in a supine position.
  * The intercostals pace is opened .
  * Chest tube is inserted in proper position regarding the site of fluid collection.
  Interventions: Procedure: Tube thoracostomy

INTERVENTIONS:
Procedure: Uniportal VATS — * single port video-assisted thoracoscopic surgery in the 5th intercostal space
  * performed under general anesthesia.
  * pleural fluid/pus was drained
  * pleural adhesions was removed
  Arms: 1
Procedure: Tube thoracostomy — * Chest tube is inserted in 5th mid-axillary line
  * performed under local anaesthesia
  Other Names: Chest tube
  Arms: 2

SUMMARY:
This randomized controlled study compared uniportal video-assisted thoracoscopic surgery (U-VATS) versus chest tube drainage for initial (first-line) treatment of stage I (exudative) and stage II (fibrinopurulent) empyema in adult patients (>18 years old). The primary end-point of outcome was the overall success of treatment (no need for re-intervention or death). The main results demonstrated the safety of minimally invasive U-VATS procedure in the initial treatment of early stages of pleural empyema in comparison to traditional chest tube drainage. Initial use of U-VATS was safe and feasible due to postoperative freedom from complex or marked effusion, in addition to significant reduction in the need for additional intervention, postoperative complications, length of hospital stay, and total cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have empyema and indicated for surgery.
* Age above 18 years old

Exclusion Criteria:

* Inability to tolerate single lung ventilation.
* Contraindication for general anesthesia/ medically unfit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Need for further management | 6 months after inital treatment
  Need for further method for pleural fluid drainage or decortication.
Mortality | 6 months after inital treatment
  Postoperative in-hospital or follow-up death.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M Elsayed, MD, Principal Investigator — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No